CLINICAL TRIAL: NCT05081687
Title: A Prospective Randomized Controlled Trial of Total Neo-adjuvant Therapy vs Conventional Chemo-radiation Aiming at Increasing Rates of Clinical Complete Response in Locally Advanced Rectal Cancer
Brief Title: Brazilian Total Neoadjuvant Therapy Trial
Acronym: BRAZIL-TNT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4015-20
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Neoplasms
Keywords: Rectal cancer; Neoadjuvant chemo-radiation; Total neoadjuvant therapy; Watch-and-wait
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — folfirinox; FOLFOXIRI protocol; Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to one of two arms: TNT and conventional therapy (control). Randomization will be stratified by study site and tumor stage (II vs III)
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total neoadjuvant therapy (TNT) (Experimental): 4 cycles of mFOLFIRINOX every 14 days:
  * Oxaliplatin 85 mg/m2
  * Irinotecan 150mg/m2
  * 5-FU 2.400mg/m2
  * Dexamethasone 12mg
  * Atropine 0.5mg
  * Netupitant/palonosetron
  Interventions: Drug: Folfirinox
- Standard of care (No Intervention): Standard post-radiation care

INTERVENTIONS:
Drug: Folfirinox — 5-FU 2400mg/m2; Oxaliplatin 85 mg/m2, Irinotecan 150mg/m2
  Other Names: mFOLFIRINOX; FOLFOXIRI; 5-FU, oxaliplatin, irinotecan
  Arms: Total neoadjuvant therapy (TNT)

SUMMARY:
Standard therapy for localized rectal cancer includes chemotherapy and radiation therapy, followed by a "recovery" period of 7-12 weeks, surgery and adjuvant chemotherapy for 3-6 months. Even though this protocol achieves high cure rates, many patients need a rectal amputation with placement of definitive colostomies. About 10-20% of patients have a complete clinical response to chemo-radiation and no tumor can be found in the surgical specimen. These patients can be followed with close surveillance and avid surgery. The aim of this study is to evaluate if a strategy including the use of a highly active chemotherapy called "FOLFIRINOX" during the 12 weeks between the end of radiation therapy and evaluation for surgery increases the rates of complete response and, therefore, allows more patients to undergo non-surgical management.

DETAILED DESCRIPTION:
Adult patients with locally advanced rectal cancer who have completed conventional long-course chemo-radiation of 54Gy with capecitabine will be randomized 1:1 to a total neo-adjuvant therapy (TNT) protocol or to a control group. Patients in the TNT arm will receive 4 cycles of interval chemotherapy with FOLFIRINOX (5-FU, irinotecan, oxaliplatin) between the end of chemo-radiation and re-staging and those in the control group will undergo standard post-radiation care during this period. All patients will be re-staged with colonoscopy and pelvic MRI 12 weeks after the end of chemo-radiation. Those with a complete clinical response will be placed under a watch-and-wait protocol with digital rectal examinations every 2 months and pelvic MRI and sigmoidoscopy every 6 months. Those wih residual tumors will undergo resection with total mesorectal excision (TME). Patients with a "near complete response", as defined by a multidisciplinary tumor board, will be re-staged at week 16 or 18 after chemo-radiation before undergoing surgery. Adjuvant chemotherapy will be done following the local standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 y/o
* Biopsy-confirmed rectal adenocarcinoma
* Tumor Stage T3+ or N+ M0
* Adequate liver function (total bilirubin < = 4.0)
* Adequate kidney function (calculate creatinine-clearance >=30ml/m2/min)
* Adequate bone marrow function (Platelet counts >=90.000, hemoglobin >=8mg/dl, neutrophile count >= 1.500/cm3)
* Completed chemo-radiation with at least 54Gy and capecitabine 1650mg/m2/d

Exclusion Criteria:

* Prior tumor resection
* Prior radiation to the pelvis
* Prior chemotherapy for rectal cancer
* Life expectancy < 6 months
* Unfit for surgery
* Need for urgent/ immediate surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
cCR + PathCR | 12 weeks after the end of chemoradiation
  Complete clinical response or pathological response

SECONDARY OUTCOMES:
Rate of R0 resection | 12 weeks
  Rate of tumor resection with negative margins
Rate of organ preservation | 6 months after surgery
  Rate of patients who remain colostomy-free
Overall toxicity | 12 weeks
  Grade 3-4 toxicities according to CTCAE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Diogo Gomes, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Municipal Vila Santa Catarina, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Program of the Brazilian Ministry of Health that us sponsoring the trial — https://hospitais.proadi-sus.org.br/